CLINICAL TRIAL: NCT05959434
Title: Integration of Cognitive Processing Therapy and Relapse Prevention for Alcohol Use Disorder and Co-Occurring PTSD: A Randomized Clinical Trial
Brief Title: Integration of Cognitive Processing Therapy and Relapse Prevention for Alcohol Use Disorder and PTSD
Acronym: CPT+RP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Medical University of South Carolina (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anka Vujanovic, Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2023-0985 / 162260; R01AA030157 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-07-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder; Alcohol Use Disorder
Keywords: trauma or PTSD; alcohol use; Cognitive Processing Therapy; Relapse Prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Wounds and Injuries; Alcohol Drinking | interventions — Secondary Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Cognitive Processing Therapy and Relapse Prevention (CPT+RP) (Experimental): Participants will receive 12, 90-minute individual sessions of CPT+RP delivered twice-weekly. We will offer some flexibility (e.g., due to illness or scheduling conflicts) and allow up to 9 weeks to complete all 12 sessions if needed. During CPT+RP, patients receive psychoeducation pertaining to the interconnectedness of AUD and PTSD and learn techniques to identify and manage triggers for alcohol use, cope with cravings, address problem thoughts about drinking, and enhance social support. These skills address core functional outcomes relevant to addiction, including executive functioning, incentive salience, and negative emotionality. The PTSD treatment component of CPT+RP reduces PTSD symptoms via identifying and targeting maladaptive trauma-related cognitions, beliefs, and Stuck Points via cognitive restructuring exercises, such as Socratic questioning. RP skills are integrated within each session.
  Interventions: Behavioral: Cognitive Processing Therapy + Relapse Prevention
- Relapse Prevention (RP) (Active Comparator): Participants will receive 12, 90-minute individual sessions of RP delivered twice-weekly as consistent with the experimental condition. The RP manual is adapted from the NIAAA Project MATCH Cognitive-Behavioral Coping Skills Therapy Manual and has been used in prior NIH-funded trials of integrated, trauma-focused treatment. Session topics include, for example, Triggers for Alcohol Use, Coping with Cravings and Urges to Drink (e.g., avoid alcohol cues, distracting activities, talk to friends/family, urge surfing), Managing Thoughts about Alcohol and Drinking by challenging and changing thoughts, Planning for Emergencies and Coping with a Lapse, Drink Refusal Skills, Increasing Pleasant Activities and Enhancing Social Support.
  Interventions: Behavioral: Relapse Prevention

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy + Relapse Prevention — Cognitive-Behavioral Therapy that integrates Cognitive Processing Therapy for PTSD with Relapse Prevention for alcohol use disorder
  Arms: Integrated Cognitive Processing Therapy and Relapse Prevention (CPT+RP)
Behavioral: Relapse Prevention — Cognitive-Behavioral Therapy that targets alcohol use, specifically
  Arms: Relapse Prevention (RP)

SUMMARY:
The goal of this clinical trial is to test the efficacy of a novel integrative cognitive-behavioral intervention in patients with posttraumatic stress disorder (PTSD) and alcohol use disorder (AUD).

Specific Aim 1: Examine the efficacy of CPT-RP, as compared to RP alone, in reducing alcohol frequency (percent days drinking) and quantity (drinks per drinking day) as measured by the Timeline Follow-Back (TLFB).

Specific Aim 2: Examine the efficacy of CPT-RP, as compared to RP alone, in reducing PTSD symptoms as measured by the Clinician Administered PTSD Scale (CAPS-5).

Specific Aim 3: Use ecological momentary assessment (EMA) to evaluate intervention effects on daily alcohol-related cognitions and behaviors through real-time associations with PTSD symptomatology and distress tolerance.

Researchers will compare integrative CPT+RP with RP-alone to see if CPT+RP is more efficacious in reducing alcohol use and PTSD symptom severity.

DETAILED DESCRIPTION:
A substantial proportion of individuals with alcohol use disorder (AUD) also meet criteria for posttraumatic stress disorder (PTSD). The co-occurrence of AUD/PTSD is characterized by more severe symptomatology, greater functional impairment, increased suicide risk, and poorer treatment outcomes as compared to either disorder alone. Trauma-focused, cognitive-behavioral interventions delivered alongside interventions for substance use disorders are most effective in reducing PTSD severity and substance use. Cognitive Processing Therapy (CPT) for PTSD and Relapse Prevention (RP) for AUD are two of the most widely used and efficacious behavioral treatments for these conditions. The investigators successfully developed and pilot tested a therapy manual that combines CPT with RP. The preliminary data demonstrate safety, feasibility, high rates of retention (80.0%) and patient satisfaction. Moreover, our data from a recent national survey of frontline mental health providers indicate that CPT is the most commonly used trauma-focused treatment for PTSD and providers are highly interested in an integrative CPT-RP intervention, conferring strong potential for uptake in real-world practice settings. In fact, due to the lack of an available, empirically developed, manualized CPT-RP treatment, 84.0% of frontline providers report attempting on their own to create such a treatment to use with their patients. This may result in highly variable and suboptimal implementation and outcomes. In response to provider input and positive preliminary data, the proposed study directly addresses this critical need by evaluating a new integrative CPT-RP treatment for individuals with co-occurring AUD and PTSD. At present, only one trauma-focused, integrative intervention is available for AUD/PTSD and it uses Prolonged Exposure (PE) to reduce PTSD symptoms. In comparison to PE, CPT is more widely used, often preferred by clinicians, equally as effective in reducing PTSD symptoms, and associated with lower dropout rates. Thus, the new CPT-RP intervention could have wider reach and greater acceptability than exposure-based treatments. Treatment choice is related to improved treatment outcomes, and therefore, there is an immediate need to add to the portfolio of evidence-based, trauma-focused, integrative treatments for AUD/PTSD. The primary objective of this Stage II study is to examine the efficacy of CPT-RP, as compared to RP alone, in reducing (1) alcohol use frequency and quantity and (2) PTSD symptom severity among individuals with current AUD/PTSD. To accomplish this, a randomized study design, manualized intervention, and standardized repeated dependent measures of clinical outcomes at multiple time points will be employed. Putative mechanisms of behavior change will be evaluated via daily monitoring. The proposed study aligns closely with the mission of NIAAA in that it aims to produce maximally efficacious behavioral interventions for AUD and comorbid psychiatric disorders such as PTSD. The findings from this study will provide new information to advance the science of AUD/PTSD comorbidity and innovate clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender identity, any race or ethnicity, aged 18-70 years.
2. Able to provide written informed consent.
3. Ability to understand English.
4. Meet DSM-5 diagnostic criteria for current (past month) moderate to severe alcohol use disorder ( >= 4 criteria).
5. At least 3 to 4 heavy drinking days per week (4 or more drinks for a woman, 5 or more drinks for a man) in the last 30 days, or >14 drinks per week for females or > 21 drinks per week for males for at least 2 weeks in the last 30 days.
6. Meet DSM-5 diagnostic criteria for current (past month) PTSD as assessed by the CAPS-5.
7. Participants may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or anxiety disorders. The inclusion of participants with affective and anxiety disorders is essential because of the marked frequency of the co-existence of mood and anxiety disorders among patients with AUD and PTSD. Concurrent substance use disorders are acceptable provided alcohol is the participant's primary substance of choice.
8. Participants taking psychotropic medications will be required to be maintained on a stable dose for at least 4 weeks before study initiation.

Exclusion Criteria:

1. Meeting DSM-5 criteria for a history of or current psychotic disorder or bipolar disorder, or imminent risk of suicidal or homicidal behavior. The intervention may be insufficient, and those participants will be referred clinically for a higher level of care.
2. Participants on psychotropic medications which have been initiated during the past 4 weeks.
3. Acute alcohol withdrawal as indicated by CIWA-Ar scores >8. Those participants will be referred clinically for medically supervised detoxification. They may be re-evaluated for eligibility after detoxification.
4. Pregnancy or breastfeeding for women.
5. Currently enrolled in evidence-based behavioral treatment for AUD or PTSD. Attendance at therapeutic activities (e.g., Alcoholics Anonymous) other than study sessions will be closely monitored using the Treatment Services Review.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use | through study treatment completion, an average of 12 weeks
  Composite of alcohol use frequency (percent days drinking) and quantity (drinks per drinking day), as measured by the Timeline Follow-Back
Change in Posttraumatic Stress Disorder (PTSD) Symptoms | through study treatment completion, an average of 12 weeks
  PTSD symptoms as measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5)

SECONDARY OUTCOMES:
Change in Alcohol Use | At 3 months, 6 months, and 12 months following study treatment completion
  Composite of alcohol use frequency (percent days drinking) and quantity (drinks per drinking day), as measured by the Timeline Follow-Back
Change in Posttraumatic Stress Disorder (PTSD) Symptoms | At 3 months, 6 months, and 12 months following study treatment completion
  PTSD symptoms as measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5)

CONTACTS AND LOCATIONS:
Overall Officials: Anka A Vujanovic, Ph.D., Principal Investigator — Texas A&M University; Sudie E Back, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas A&M University, College Station, Texas

IPD SHARING:
Plan to Share IPD: Yes